CLINICAL TRIAL: NCT04804228
Title: Comparison of the Efficacy of Electrical Dry Needling Versus Traditional Physical Therapy in the Treatment of Active Myofascial Trigger Points in Pain, Sensitivity, Functionality and Quality of Life of Patients With Chronic Non-specific Low Back Pain
Brief Title: Efficacy of Electrical Dry Needling in Pain, Sensitivity, Functionality and Quality of Life of Patients With Chronic Non-specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Responsible Party: Principal Investigator, Adelaida María Castro-Sánchez, Principal Investigator, Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFM 87/2020
Record Dates: First submitted 2021-01-14; First posted 2021-03-18 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-11

CONDITIONS: Chronic Low-back Pain
Keywords: Electrical dry needling; low back pain; Randomized clinical trial; ischemic compression; analytical stretch
MeSH Terms: conditions — Low Back Pain | interventions — Acupressure

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electrical dry needling (Experimental): The experimental group consisting of 40 subjects will perform electrostimulation on the active myofascial trigger points of the following muscles: quadratus lumbar, multifidus and iliocostalis, following the PGM maps described by Travell and Simons. The electrostimulation of the PGM will be carried out using needle electrodes, the generated current will be produced by a TENS device with a frequency of 2 Hz and a pulse width of 250 μs, the application will be approximately 30 min. The therapeutic intervention will be 1 session per week for a total of 6 weeks.
  Interventions: Other: Ischemic compression, analytical stretching and postural habits educational dossier
- Ischemic compression, analytical stretching and postural habits educational dossier (Active Comparator): The control group consisting of 40 subjects will undergo an ischemic compression technique in active PGM with a time between 20 seconds and 1 minute until pain inhibition is achieved, and finally, analytical stretching will be carried out on the quadratus lumbar, multifid and iliocostal, 1 weekly session for 6 weeks providing a training dossier of postural education in their activities of daily life.
  Interventions: Other: Electrical dry needling

INTERVENTIONS:
Other: Electrical dry needling — The experimental group consisting of 40 subjects will perform electrostimulation on the active myofascial trigger points of the following muscles: quadratus lumbar, multifidus and iliocostalis. The electrostimulation of the PGM will be carried out using needle electrodes, the generated current will be produced by a TENS device with a frequency of 2 Hz and a pulse width of 250 μs, the application will be approximately 30 min. The therapeutic intervention will be 1 session per week for a total of 6 weeks.
  Arms: Ischemic compression, analytical stretching and postural habits educational dossier
Other: Ischemic compression, analytical stretching and postural habits educational dossier — The control group G2, formed by 40 subjects, will perform an ischemic compression technique in active PGM with a time between 20 seconds and 1 minute until pain inhibition is achieved, and finally, analytical stretching will be carried out on the quadratus lumbar, multifidus and iliocostal muscles, 1 weekly session for 6 weeks, in addition to providing them with a training dossier on postural education in their activities of daily life.
  Arms: Electrical dry needling

SUMMARY:
The main objective of this study is to determine the efficacy of electrical dry needling versus ischemic compression, analytical stretching and postural habits educational dossier in active myofascial trigger points in patients with chronic non-specific low back pain.

DETAILED DESCRIPTION:
A double-blind clinical trial will be developed in a sample of 80 subjects with chronic low back pain. Patients in the experimental group will receive electrical dry needling at the active myofascial trigger points (PGM) of the quadratus lumbar, multifidus, and iliocostal muscles (following the PGM maps described by Travell and Simons). The technique will be performed using needle electrodes, the generated current will be produced by a TENS device with a frequency of 2 Hz and a pulse width of 250 μs, during 30 min of application. The therapeutic intervention will be 1 weekly session for a total of 6 weeks.

The control group will perform an ischemic compression technique in active PGM with a time between 20 seconds and 1 minute until pain inhibition is achieved, and finally, analytical stretching will be carried out on the quadratus lumbar, multifidus and iliocostal muscles. The treatment will consist of 1 weekly session for 6 weeks, in addition they will be provided with a training dossier on postural education in their activities of daily life.

A baseline assessment of the primary and secondary outcome measures will be carried out before randomization of the participants to the different groups, an immediate post-treatment assessment (1 day after the last intervention) and an assessment two month after the end of the intervention ( short-term follow-up).

The objectives of this study are to compare the repercussions of dry electropuncture versus ischemic compression in active PGM plus stretching in terms of pain, functionality, mobility of the spine, and quality of life in patients with non-specific chronic low back pain; and analyze the impact on active myofascial trigger points in terms of pressure tolerance threshold.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain ≥ 3 months.
* Age between 30 and 67 years old.
* Not being receiving physical therapy.

Exclusion Criteria:

* Presence of lumbar stenosis.
* Diagnosis of spondylolisthesis.
* Diagnosis of fibromyalgia.
* Treatment with corticosteroids or oral medication in recent weeks.
* History of spine surgery.
* Contraindication of analgesic electrical therapy.
* Have previously received a treatment of electrical analgesia or exercise.
* Central or peripheral nervous system disease.

Ages: 30 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-05-17 (Actual); Primary Completion 2021-08-17 (Actual); Study Completion 2021-11-20 (Actual)

PRIMARY OUTCOMES:
Changes in pressure pain threshold by Wagner manual pressure algometer. | At baseline, at 6 weeks and at 2 months
  Apply the tip of the algometer perpendicular to the muscle and maintain a pressure, which will gradually increase to 1 kg / sec. Subjects will be instructed to signal the moment they experience pain, in order to have an accurate record (pain threshold).
Change from baseline in Roland Morris Disability Questionnaire (RMDQ). | At baseline, at 6 weeks and at 2 months
  This is a self-reported questionnaire consisting in 24 items reflecting limitations in different activities of daily living attributed to low back pain including walking, vending over, sitting, lying down, dressing, sleeping, self-care and daily activities.Ranging from 0 points- better to 24 points- worse disability

SECONDARY OUTCOMES:
Change from baselina in range of motion | At baseline, at 6 weeks and at 2 months
  This variable is quantified using the SpinalMouse ® device (Phisiotech, Spain). It is an electronic computer-aided measuring device that measures sagittal spinal amplitude of movement (ROM) and intersegmental angles in a non-invasive way.
Change from baseline in lumbar mobility flexion. | At baseline, at 6 weeks and at 2 months
  For the quantification of lumbar flexion an angular inclinometer is used (Fleximeter UM 8320-3 RJ Code Research Institute, Brazil).
Changes in pressure pain threshold by Wagner manual pressure algometer. | At baseline, at 6 weeks and at 2 months
  Apply the tip of the algometer perpendicular to the muscle and maintain a pressure, which will gradually increase to 1 kg / sec. Subjects will be instructed to signal the moment they experience pain, in order to have an accurate record (pain threshold).
Tampa Scale of Kinesiophobia (TSK).Change from baseline in Fear of Movement. | At baseline, at 6 weeks and at 2 months
  Is a 17-item questionnaire that measures the fear of movement and (re)injury.Patient rate beliefs about their pain on a 4-point scale ranging from strongly disagree to strongly agree (ranging from 17-68 points).
SF-36 Health Questionnaire (SF-36).Change from baseline on Quality of Life. | At baseline, at 6 weeks and at 2 months
  The SF-36 quality of life questionnaire assesses 8 domains including physical functioning, physical role, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. This scale ranges from 0 (lowest level of functioning) to 100 (highest level)
Change from Mcquade Test. | At baseline, at 6 weeks and at 2 months
  It measures the isometric endurance of trunk flexion muscles.
Change from insomnia Severity Index Índice de calidad de sueño de Pittsburgh. | At baseline, at 6 weeks and at 2 months
  This questionnaire consists of 24 questions. The total score can range from 0 to 21 points. The higher the total score, the worse the quality of sleep.
Change from baseline in disability. Oswestry Low Back Pain Disability Idex. | At baseline, at 6 weeks and at 2 months
  It has 10 items associated to activities of daily living, each ítem has a puntuation fron 0 to 5 points.The higher scores mean a worse outcome.
Change from baseline in pain intensity. Visual analogue scale | At baseline, at 6 weeks and at 2 months
  A 10-point Numerical Pain Scale (0: no pain, 10: maximum pain) assesses the intensity of pain. Range from no pain 0 to maximum pain 10 points

CONTACTS AND LOCATIONS:
Overall Officials: Adelaida María Castro-Sánchez, PhD, Principal Investigator — Almeria University
Locations (1):
- Adelaida María Castro-Sánchez, Almería, Spain

REFERENCES:
- [Background] Chiarotto A, Clijsen R, Fernandez-de-Las-Penas C, Barbero M. Prevalence of Myofascial Trigger Points in Spinal Disorders: A Systematic Review and Meta-Analysis. Arch Phys Med Rehabil. 2016 Feb;97(2):316-37. doi: 10.1016/j.apmr.2015.09.021. Epub 2015 Oct 17. PMID 26475933
- [Background] Travell JG, Simons DG, Simons LS. Dolor y disfunción miofascial. El manual de los puntos gatillo. Volumen I. Mitad superior del cuerpo. Madrid: Ed Panamericana. 2007.
- [Background] Travell JG, Simons DG. Dolor y disfunción miofascial. El manual de los puntos gatillo. Volumen II. Extremidades inferiores. Madrid: Ed Panamericana. 2007.
- [Background] Dunning J, Butts R, Young I, Mourad F, Galante V, Bliton P, Tanner M, Fernandez-de-Las-Penas C. Periosteal Electrical Dry Needling as an Adjunct to Exercise and Manual Therapy for Knee Osteoarthritis: A Multicenter Randomized Clinical Trial. Clin J Pain. 2018 Dec;34(12):1149-1158. doi: 10.1097/AJP.0000000000000634. PMID 29864043
- [Background] Dunning J, Butts R, Henry N, Mourad F, Brannon A, Rodriguez H, Young I, Arias-Buria JL, Fernandez-de-Las-Penas C. Electrical dry needling as an adjunct to exercise, manual therapy and ultrasound for plantar fasciitis: A multi-center randomized clinical trial. PLoS One. 2018 Oct 31;13(10):e0205405. doi: 10.1371/journal.pone.0205405. eCollection 2018. PMID 30379937
- [Background] Fernandez-de-Las-Penas C, Nijs J. Trigger point dry needling for the treatment of myofascial pain syndrome: current perspectives within a pain neuroscience paradigm. J Pain Res. 2019 Jun 18;12:1899-1911. doi: 10.2147/JPR.S154728. eCollection 2019. PMID 31354339
- [Background] Rahou-El-Bachiri Y, Navarro-Santana MJ, Gomez-Chiguano GF, Cleland JA, Lopez-de-Uralde-Villanueva I, Fernandez-de-Las-Penas C, Ortega-Santiago R, Plaza-Manzano G. Effects of Trigger Point Dry Needling for the Management of Knee Pain Syndromes: A Systematic Review and Meta-Analysis. J Clin Med. 2020 Jun 29;9(7):2044. doi: 10.3390/jcm9072044. PMID 32610659
- [Background] Dunning J, Butts R, Zacharko N, Fandry K, Young I, Wheeler K, Day J, Fernandez-de-Las-Penas C. Spinal manipulation and perineural electrical dry needling in patients with cervicogenic headache: a multicenter randomized clinical trial. Spine J. 2021 Feb;21(2):284-295. doi: 10.1016/j.spinee.2020.10.008. Epub 2020 Oct 13. PMID 33065273
- [Background] Kumnerddee W, Pattapong N. Efficacy of electro-acupuncture in chronic plantar fasciitis: a randomized controlled trial. Am J Chin Med. 2012;40(6):1167-76. doi: 10.1142/S0192415X12500863. PMID 23227789
- [Background] Myburgh C, Larsen AH, Hartvigsen J. A systematic, critical review of manual palpation for identifying myofascial trigger points: evidence and clinical significance. Arch Phys Med Rehabil. 2008 Jun;89(6):1169-76. doi: 10.1016/j.apmr.2007.12.033. PMID 18503816
- [Derived] Lara-Palomo IC, Antequera-Soler E, Fernandez-Sanchez M, Castro-Sanchez AM, Garcia-Lopez H. Electrical dry needling versus a non-invasive multicomponent intervention in the treatment of myofascial trigger points in patients with chronic low back pain: A randomised clinical trial. Clin Rehabil. 2024 Mar;38(3):347-360. doi: 10.1177/02692155231201589. Epub 2023 Sep 13. PMID 37700695
- [Derived] Lara-Palomo IC, Gil-Martinez E, Antequera-Soler E, Castro-Sanchez AM, Fernandez-Sanchez M, Garcia-Lopez H. Electrical dry needling versus conventional physiotherapy in the treatment of active and latent myofascial trigger points in patients with nonspecific chronic low back pain. Trials. 2022 Mar 28;23(1):238. doi: 10.1186/s13063-022-06179-y. PMID 35346331